CLINICAL TRIAL: NCT01031667
Title: Synergistic Effect of Combination Therapy With Cilostazol and Probucol on Plaque Stabilization and Lesion Regression: Serial Intravascular Ultrasound and Virtual Histology Study(SECURE Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Won-Heum Shim / Professor of Cardiology at Severance Cardiovascular Hospital, Yonsei University Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2009-0489
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Therapy
Keywords: Patients treated with PCI with stent
MeSH Terms: interventions — Cilostazol; Probucol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cilostazol, Probucol / placebo of probucol — An investigator-initiated, placebo-controlled, randomized, multi-center study. Enrolled patients will be randomized after PCI either to the combination therapy group or to the control group. In the combination therapy group, cilostazol 200 mg and probucol 500 mg will be administered daily, whereas the control group will receive cilostazol 200 mg daily only.

SUMMARY:
The purpose of this study is to evaluate the effect of combination therapy with cilostazol and probucol on plaque volume and composition change in comparison with cilostazol alone by serial intravascular ultrasound and virtual histology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated with PCI with stent
2. Male or female over 20 years of age
3. Presence of at least one PCI target lesion(lesion length ≤26mm) with ≥50% diameter stenosis that can be covered with a single Endeavor Sprint stent(Medtronic)
4. Other PCI target lesions also should be treated with Endeavor Sprint stents
5. Presence of an intermediate non-PCI target lesion with luminal narrowing of ≥30% and ≤70% by visual estimation
6. Signed written informed consent to participate in the study

Exclusion Criteria:

1. Intermediate (non-PCI target) lesions that might provide difficulty for IVUS evaluation because of following reasons: heavy calcification (>90° Arc), tortuous vessel with sever angulation, total occlusion, or bifurcation lesions
2. Previous PCI in the last 6 months
3. Previous CABG
4. Patients with AMI undergoing primary PCI or rescue PCI after thrombolysis
5. Cardiogenic shock
6. Inability to take adequate anti-platelet therapy
7. Thrombocytopenia (platelet count <70 x 109/l)
8. Known hypersensitivity or contraindication to any of the following medications: Heparin, aspirin, clopidogrel, cilostazol, probucol, statin, contrast media*

   *Patients with documented sensitivity to contrast media which can be effectively pre-medicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Those with true anaphylaxis to prior contrast media, however, should not be enrolled.
9. History of severe ventricular arrhythmia
10. Significant QTc prolongation (≥470 ms) on ECG
11. NYHA class III/IV heart failure or LV ejection fraction ≤35%
12. Familial hypercholesterolemia
13. Uncontrolled hypertriglyceridemia (>400 mg/dL)
14. Chronic renal failure with serum creatinine level ≥2mg/dL
15. Severe liver disease or transaminase level ≥3 times the upper limit of normal.
16. Pregnant or breastfeeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Plaque volume change of the index lesion with intermediate stenosis(non-PCI target lesion) | From February 01, 2009 to July 31, 2011

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

REFERENCES:
- [Derived] Ko YG, Kim BK, Lee BK, Kang WC, Choi SH, Kim SW, Lee JH, Lee M, Honda Y, Fitzerald PJ, Shim WH; SECURE Investigators. Study design and rationale of "Synergistic effect of combination therapy with cilostazol and ProbUcol on plaque stabilization and lesion REgression (SECURE)" study: a double-blind randomised controlled multicenter clinical trial. Trials. 2011 Jan 12;12:10. doi: 10.1186/1745-6215-12-10. PMID 21226953